CLINICAL TRIAL: NCT05576272
Title: A Randomized, Open, Multicenter Phase II/III Trial to Compare the Efficacy and Safety of QL1706 and Carrilizumab Combined With Gemcitabine and Cisplatin in First-line Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: A Phase II/III Trial to Evaluate the Efficacy and Safety of QL1706 in Patients With Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-302
Record Dates: First submitted 2022-09-30; First posted 2022-10-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 Combined with Gemcitabine and Cisplatin (Experimental)
  Interventions: Drug: QL1706; Drug: Gemcitabine; Drug: Cisplatin
- Carrilizumab Combined with Gemcitabine and Cisplatin (Active Comparator)
  Interventions: Drug: Carrelizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: QL1706 — 5 mg/kg#D1#Q3W IV, 4-6 cycles
  Arms: QL1706 Combined with Gemcitabine and Cisplatin
Drug: Carrelizumab — 200mg#D1#Q3W IV, 4-6 cycles
  Arms: Carrilizumab Combined with Gemcitabine and Cisplatin
Drug: Gemcitabine — 1000mg/m2#D1&D8#Q3W IV, 4-6 cycles
Drug: Cisplatin — 80mg/m2#D1#Q3W IV, 4-6 cycles

SUMMARY:
This is a randomized, open, multicenter phase II/III trial to compare the efficacy and safety of QL1706 and carrilizumab combined with gemcitabine and cisplatin in first-line treatment of recurrent or metastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a randomized, open, multicenter phase II/III trial to compare the efficacy and safety of QL1706 and carrilizumab combined with gemcitabine and cisplatin in first-line treatment of recurrent or metastatic nasopharyngeal carcinoma. The study is divided into two parts.

The first part is a phase II, single-arm study with an introductory safety phase, which is planned to enroll 30 subjects with nasopharyngeal carcinoma treated with first-line QL1706 in combination with gemcitabine and cisplatin. The primary objective of the first part is to evaluate the safety and tolerability of QL1706 combined with gemcitabine and cisplatin in the first-line treatment of patients with recurrent or metastatic nasopharyngeal carcinoma.

The second part is a phase III randomized, controlled study. The study plans to enroll 430 subjects, who will be randomized in a 1:1 ratio to a trial group of QL1706 in combination with gemcitabine and cisplatin and a control group of carrilizumab in combination with gemcitabine and cisplatin. The primary objective of the second part was to compare the effectiveness of QL1706 with that of carrilizumab combined with gemcitabine and cisplatin, respectively, in the first-line treatment of recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The subject will participate voluntarily and sign the informed consent form.
2. Age ≥ 18 years when signing the informed consent form, male or female.
3. The Eastern Collaborative Oncology Group (ECOG) physical status score was 0 or 1.
4. Expected survival ≥ 3 months.
5. Patients with pathologically confirmed nasopharyngeal carcinoma.
6. Patients with primary diagnosis of metastatic nasopharyngeal carcinoma [stage IVb according to the American Joint Committee on Cancer AJCC staging system (8th edition)] or patients with recurrent (including recurrent or metastatic) nasopharyngeal carcinoma who are not candidates for radical surgery or radiotherapy or other local treatment; and for recurrent or metastatic lesions must be untreated systemically: previously treated with neoadjuvant chemotherapy with curative intent, Patients with adjuvant chemotherapy, radiotherapy or radiotherapy must have had ≥ 6 months between the last chemotherapy and or radiotherapy and the time of disease recurrence and/or development of metastases.
7. Patients have at least one imaging measurable lesion according to RECISTv1.1 evaluation criteria; for lesions that have received prior radiotherapy or other local treatment there must be evidence of definite progression of the lesion after the end of local treatment in order to be selected as a measurable lesion.
8. Adequate organ function prior to first use of the experimental drug (no blood components, leukocyte-raising drugs, or platelet-raising drugs are allowed within 7 days prior to obtaining laboratory tests)

   1. Absolute neutrophil count ≥ 1.5 x 109/L.
   2. Platelet count ≥ 100×109/L.
   3. Hemoglobin ≥ 90 g/L.
   4. Serum albumin ≥ 28 g/L.
9. Subjects (both female and male) agree to use effective contraception from the time they sign the informed consent until 180 days after the last use of the trial drug. Women who are not pregnant or breastfeeding from the time they sign informed consent until 180 days after the last use of the trial drug.

Exclusion Criteria:

1. Presence of symptomatic central nervous system (CNS) metastases, soft meningeal metastases, or spinal cord compression due to metastases.
2. Prior systemic anticancer treatment with approved drugs or trial drugs.
3. End date of palliative radiotherapy targeting bone metastases or soft tissue, etc. ≤ 7 days from imaging of baseline tumor lesions
4. Presence of carcinomatous meningitis prior to first study treatment
5. Active autoimmune disease present within 2 years prior to the first administration of the investigational drug and requiring systemic systemic therapy. Subjects with relevant alternative therapy who are stable are allowed to be included.
6. Disease requiring systemic treatment with corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive drugs present within 2 weeks prior to first study treatment.
7. At the investigator's discretion, have a serious concomitant condition that jeopardizes patient safety, or interferes with patient completion of the study, such as hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) not controlled by two or more antihypertensive medications, or severe diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) -BICR | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months after the last QL1706 injection has been administered
  The PFS assessed by Blinded independent central review (BICR)

SECONDARY OUTCOMES:
PFS- Investigator | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months after the last QL1706 injection has been administered
  The PFS assessed by Investigator
Objective remission rate (ORR) | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 72 weeks
  The ORR assessed by BICR and Investigator
Duration of remission (DOR) | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 72 weeks
  The DOR assessed by BICR and Investigator
Disease Control Rate (DCR) | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 72 weeks
  The DCR assessed by BICR and Investigator
Overall survival (OS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months after the last QL1706 injection has been administered
  Overall survival
12-month OS rate | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months after the last QL1706 injection has been administered
  12-month Overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: li Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No